CLINICAL TRIAL: NCT06854887
Title: The Added Value of Digital Breast Tomosynthesis Over Mammography in Local Tumor Staging in Patients With BIRADS 4 or 5 Lesions
Brief Title: The Added Value of DBT Over Mammography in Local Tumor Staging in Patients With BIRADS 4 or 5 Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Silvia Gamal Rasmy, resident doctor, Assiut University
Other Study IDs: DBT &Mammography in BIRADS 4-5
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Digital Breast Tomosynthesis
MeSH Terms: interventions — Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: digital breast tomosynthesis and mammography — tomosynthesis is 3D image for the breast mammography is 2D image for the breast

SUMMARY:
Compare the diagnostic accuracy of tomosynthesis with 2D mammography in cases with suspected BI-RADS 4 or 5 to determine its potential benefit for staging

DETAILED DESCRIPTION:
Digital breast tomosynthesis (DBT) is a promising 3D imaging technique for breast imaging that use in breast cancer detection. it acquires reconstructed volume data , the data is reconstructed secondarily in mammary slices from several radiographs acquired from different angles of view (-15◦ to +15◦ for Fuji). It theoretically improves the sensitivity of detection by enabling enhanced delimitation of the lesion margins, and the specificity by avoiding the problem of glandular superimposition, By separating overlapping breast tissues & it enhances detection of abnormalities located in different planes. DBT has higher breast cancer detection rates and lower recall rates compared with digital mammography (DM). There is also evidence of the diagnostic efficacy of DBT in women with clinical symptoms and women with screen-detected findings who have been recalled for work-up. Consequently, recommendations have been made about the role of DBT in screening asymptomatic women according to their risk levels, in evaluation of symptomatic women, and in work-up of suspicious DM findings. The main objective of this study was to compare tomosynthesis with 2D mammography in cases with suspected BI-RADS 4 or 5 anomalies, to determine its potential benefit for staging.

ELIGIBILITY:
Inclusion Criteria:

1. BI-RADS 4 OR 5 LESION that pathologically proved to be breast cancer.
2. No history of previous operations
3. No history of chemotherapy or radiotherapy

Exclusion Criteria:

1. BI-RADS 1 ,2,3 lesions
2. History of previous operation

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study included patients with BIRADS 4 or 5 lesions who pathologically proved to be breast cancer by TCNB
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-03-29 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Recording The breast density in both tomosynthesis and mammography for the main and satellite lesions | baseline
  The breast density according to ACR BIRADS in both tomosynthesis and mammography for the main and satellite lesions
Recording the type of lesion in both tomosynthesis and mammography for the main and satellite lesions | baseline
  the type of lesion (mass , microcalcification , architectural distortion) in both tomosynthesis and mammography for the main and satellite lesions
Recording the probability of multifocality or multicentricity in both tomosynthesis and mammography for the main and satellite lesions | baseline
  the probability of multifocality or multicentricity in both tomosynthesis and mammography for the main and satellite lesions
Recording the location of the tumor within the mammary quadrants and the depth of the tumor in both tomosynthesis and mammography for the main and satellite lesions | baseline
  The location of the tumor within the mammary quadrants (upper , lower , outer , inner ) and the depth (anterior-middle-posterior) of the tumor in both tomosynthesis and mammography for the main and satellite lesions
Recording the tumor histopathology type for the main and satellite lesions | baseline
  Recording the tumor histopathology type (ductal, lobular , in situ , others) for the main and satellite lesions

REFERENCES:
- [Result] Mariscotti G, Durando M, Houssami N, Fasciano M, Tagliafico A, Bosco D, Casella C, Bogetti C, Bergamasco L, Fonio P, Gandini G. Comparison of synthetic mammography, reconstructed from digital breast tomosynthesis, and digital mammography: evaluation of lesion conspicuity and BI-RADS assessment categories. Breast Cancer Res Treat. 2017 Dec;166(3):765-773. doi: 10.1007/s10549-017-4458-3. Epub 2017 Aug 17. PMID 28819781
- [Result] Bernardi D, Belli P, Benelli E, Brancato B, Bucchi L, Calabrese M, Carbonaro LA, Caumo F, Cavallo-Marincola B, Clauser P, Fedato C, Frigerio A, Galli V, Giordano L, Giorgi Rossi P, Golinelli P, Morrone D, Mariscotti G, Martincich L, Montemezzi S, Naldoni C, Paduos A, Panizza P, Pediconi F, Querci F, Rizzo A, Saguatti G, Tagliafico A, Trimboli RM, Zappa M, Zuiani C, Sardanelli F. Digital breast tomosynthesis (DBT): recommendations from the Italian College of Breast Radiologists (ICBR) by the Italian Society of Medical Radiology (SIRM) and the Italian Group for Mammography Screening (GISMa). Radiol Med. 2017 Oct;122(10):723-730. doi: 10.1007/s11547-017-0769-z. Epub 2017 May 25. PMID 28540564
- [Result] Marinovich ML, Hunter KE, Macaskill P, Houssami N. Breast Cancer Screening Using Tomosynthesis or Mammography: A Meta-analysis of Cancer Detection and Recall. J Natl Cancer Inst. 2018 Sep 1;110(9):942-949. doi: 10.1093/jnci/djy121. PMID 30107542